CLINICAL TRIAL: NCT05564260
Title: The Effects of Virtual Reality and Kaleidoscope on Pain and Fear During Blood Draw in Children: A Randomized Controlled Trial
Brief Title: The Effects of Virtual Reality and Kaleidoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Esra TURAL BUYUK, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0.20.08/687-905- 10.10.2019
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Fear; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Kaleidescope Group (Experimental): Kaleidoscope was watched during blood drawing
  Interventions: Behavioral: Kaleidescope
- The VR Group (Experimental): watching the application by wearing virtual glasses to the child during the blood drawing
  Interventions: Behavioral: Virtual Reality
- Control Group (No Intervention): No intervention was made.

INTERVENTIONS:
Behavioral: Kaleidescope — watching kaleidescope
  Other Names: distraction methods
  Arms: The Kaleidescope Group
Behavioral: Virtual Reality — wearing virtual reality glasses
  Other Names: distraction methods
  Arms: The VR Group

SUMMARY:
In literature review, many studies have been found to support the positive effects of various nonpharmacological methods in the alleviation of pain and fear created by invasive procedures.This study was carried out to determine the effects of kaleidoscope and cartoon watching using the virtual reality glasses on the pain and fear states of children during blood draw procedure.

DETAILED DESCRIPTION:
This study was carried out to determine the effects of kaleidoscope and cartoon watching using the virtual reality glasses on the pain and fear states of children during blood draw procedure.

H0: There are no significant differences in the mean pain and fear scores of the children who used kaleidoscope and cartoon watching using virtual reality glasses methods.

H1: Mean pain and fear score of the children who used kaleidoscope during blood draw procedure is lower than the ones who did not.

H2: Mean pain and fear score of the children who used virtual reality glasses during blood draw procedure is lower than the ones who did not.

This study was carried out with 7-12 year old children who were admitted to blood draw unit of a hospital in Turkey between January 21-April 21, 2020. Sample size was calculated as 156 including 52 individuals per each group in the study (52 in the kaleidoscope group, 52 in the virtual reality group and 52 in the control group). However, 2 children were lost in all groups due to the inability to draw blood with one entry and data were completed with a total of 150 children. Groups were generated by using randomization method. Participant Information Form: This form included sociodemographic characteristics (age, sex, presence of chronic disease) of the children.

Visual Analog Scale (VAS): Visual Analog Scale, which is used to measure severity of pain consists of a horizontal or vertical ruler at a length of 10 cm or 100 mm which has "no pain" on one side and "the most severe pain possible" on the other side. While there is "no pain" expression on the left side of the ruler, there is "unberable pain" expression on the right side. VAS is described as understandable and easy-to-use for the children over 7 years old. Its validity and reliability have been shown in the previous studies. 14-16 Wong-Baker FACES Pain Rating Scale (FACES): This scale is used for children aged 3 years and older in order to rate severity of pain. In this numerical rating scale, scores given by the child range between 0 and 10. Faces show emotions from smiling (0= very happy/no pain) to crying (10= the most painful).17 In this study, children were assessed by the researcher and nurse in the clinic during post-procedure. Wong-Baker Faces Pain Rating Scale (FACES) is a commonly used scale to evaluate pain in pediatric group in Turkish population. 11,18 The Children's Fear Scale (CFS): This is a one-item self-report scale which is used to measure pain-associated fear. This one-item scale is composed of five neutral faces in terms of sex. There is a face showing no fear on the left and a face showing extreme fear on the right. The response of the evaluator shows the level of fear. It can be used by the parents and researchers before and during the procedure for the children aged 5-10 years old.19,20 The directions of Children's Fear Scale was changed in line with the fear-related word capacity of the children developmentally.19 Psychometric properties of the scale in Turkish population were carried out by Gerceker, Ayar, Ozdemir et al. 20 Fear scale was assessed before and after the blood draw procedure by the child, parent and researcher during the study.

'VR BOX 3D' virtual reality glasses compatible with smartphones were used in the study. While using VR, there is no need for any power or connection unit other than the phone. All children in the study were made to watch the same video (Puss in Boots The Three Musketeers/Looney Tunes Road Runner) recommended by the experts based on children ages. Five children between 7-12 years old were made to watch selected videos before starting the study. There was no negative feedback

ELIGIBILITY:
Inclusion Criteria:

* being literate for the child and parent
* being 7-12 years old
* having no vision or hearing problems
* having no chronic or mental health problem.

Exclusion Criteria:

* the child with physical and psychological deficit to prevent him from wearing the glasses to be worn on his head so that he can watch virtual reality.
* having vision or hearing problems
* having chronic or mental health problem.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 156 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Pain assesed by child, parent, nurse with Wong-Baker FACES | during procedure
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Pain assesed by Visual Analohg Scale (VAS) | during procedure
  Visual Analog Scale (VAS): Visual Analog Scale, which is used to measure severity of pain consists of a horizontal or vertical ruler at a length of 10 cm or 100 mm which has "no pain" on one side and "the most severe pain possible" on the other side. While there is "no pain" expression on the left side of the ruler, there is "unberable pain" expression on the right side. VAS is described as understandable and easy-to-use for the children over 7 years old. Its validity and reliability have been shown in the previous studies
Fear assesed by The Children's Fear Scale (CFS) | during procedure
  This is a one-item self-report scale which is used to measure pain-associated fear. This one-item scale is composed of five neutral faces in terms of sex. There is a face showing no fear on the left and a face showing extreme fear on the right. The response of the evaluator shows the level of fear. It can be used by the parents and researchers before and during the procedure for the children aged 5-10 years old

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tural Buyuk, Principal Investigator — Phd, RN
Locations (1):
- Bafra State Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No